CLINICAL TRIAL: NCT06819930
Title: Assessment of the Functional Capacity of Patients with Fibromyalgia: Clinical Validity and in the Determination of Work Incapacity
Brief Title: Assessment of the Functional Capacity of Patients with Fibromyalgia: Clinical Validity
Status: Enrolling by invitation | Type: Observational
Sponsor: University Ramon Llull (Other)
Responsible Party: Principal Investigator, Blanca Roman-Viñas, MD, PhD, University Ramon Llull
Other Study IDs: URamonLlull
Record Dates: First submitted 2025-01-22; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Fibromyalgia (FM); Work Ability; Physical Activity; Physical Functioning; Physical Performance
MeSH Terms: conditions — Fibromyalgia; Motor Activity | interventions — Surveys and Questionnaires; Accelerometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Women with Fibromyalgia who are actively working
  Interventions: Other: Physical Assessments, Questionnaires, and Accelerometry for Fibromyalgia evaluation
- Women with Fibromyalgia on sick leave
  Interventions: Other: Physical Assessments, Questionnaires, and Accelerometry for Fibromyalgia evaluation
- Women with Fibromyalgia with permanent work disability (oficially recognized by the INSS)
  Interventions: Other: Physical Assessments, Questionnaires, and Accelerometry for Fibromyalgia evaluation
- Control group of sedentary women without Fibromyalgia
  Interventions: Other: Physical Assessments, Questionnaires, and Accelerometry for Fibromyalgia evaluation

INTERVENTIONS:
Other: Physical Assessments, Questionnaires, and Accelerometry for Fibromyalgia evaluation — This study involves a combination of functional tests, questionnaires, and activity measurement using accelerometers. The functional tests include the six-minute walk test (6MWT), handgrip strength dynamometry, and the 8-foot up & go test. Participants will also complete validated questionnaires assessing symptoms, quality of life, and psychosocial impact. Additionally, accelerometers will be used to objectively measure physical activity levels throughout the study period

SUMMARY:
Fibromyalgia is one of the main causes of chronic pain without a specific etiology, affecting 8% of the Spanish population, especially women. Its most characteristic symptoms include generalized pain, fatigue, difficulty falling asleep, joint stiffness, anxiety, and depression. Due to the lack of objective data confirming the condition and the subjectivity of the symptoms, the current diagnosis is purely clinical. Moreover, despite the significant impact on the quality of life of those who suffer from it, there is a lack of scientific evidence to assess the degree to which it affects their functional and work capacity. This concept is gaining relevance in the growing context of patients seeking work disability.

Thus, due to the lack of international consensus and standardized protocols, this study hypothesizes that the functional capacity of Spanish women with fibromyalgia, aged 30 to 64, evaluated with various validated tests such as the six-minute walking test (6MWT), handgrip strength dynamometry, and the 8-foot up & go, correlates directly with their quality of life, physical activity measured by accelerometry, and social and psychological impact, provided there is no economic benefit. Therefore, the primary aim of this research is to validate a standardized protocol for evaluating the functional and work capacity of Spanish women with fibromyalgia and to assess its correlation with quality of life, physical activity, and psychosocial impact.

The study will include a total sample of 160 women, divided into four groups of 40 participants: women with fibromyalgia who are actively working, women with fibromyalgia on sick leave, women with fibromyalgia with permanent work disability (officially recognized by the National Institute of Social Security, INSS), and a control group of healthy women.

The patients will be required to attend in person to complete the full protocol, with a one-week interval between sessions. Subsequently, two follow-ups will be conducted at 6 and 12 months, where the work situation will be reassessed, and questionnaires will be administered. The protocol includes the following variables for study: age, weight, height, marital status, country of origin, socioeconomic level, educational level, occupation, work situation, generalized pain index questionnaire, symptom severity questionnaire, fibromyalgia impact questionnaire, allodynia test, six-minute walking test, 8-foot up and go, handgrip strength dynamometry, tender points, false points, SF-36 questionnaire, Hospital Anxiety and Depression Scale, multidimensional perceived social support scale, and accelerometry.

The aim of this study is to analyze in greater depth the validity of the tests currently used in clinics to objectively assess the functional capacity of patients with fibromyalgia. In this way, this study will become the first to present and evaluate the validity and reliability of a protocol for assessing functional capacity. If the proposed hypothesis is proven, these tests and evaluation methods will be highly useful for systematic incorporation into the routine of functional capacity assessment services, as well as in daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 30 and 64 years old with a diagnosis of fibromyalgia made by a rheumatologist or family doctor following the ACR diagnostic criteria.
* For the control group, women matched by age with no diagnosis of fibromyalgia and with a sedentary lifestyle will be included.
* All participants must agree to be part of the study.

Exclusion Criteria (for both case group and control group):

* Illiteracy and/or lack of understanding of Spanish.
* Severe psychiatric and/or psychological disorders, associated musculoskeletal diseases that could increase pain, such as uncontrolled endocrine disorders, autoimmune diseases, and/or other associated rheumatological or neurological conditions.
* Additionally, patients who refuse to participate in the study or any condition that, in the investigator's judgment, would prevent proper adherence to the protocol will be excluded.

Ages: 30 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will include a total of 160 women, calculated using the Epidat version 3.1 statistical software (University of Santiago de Compostela, Spain). The sample size was estimated based on the average and standard deviation of parameters considered for diagnosing fibromyalgia, the General Pain Index (IDG), and the Symptom Severity Index (EGS). The maximum acceptable error percentage is 5%, accounting for variability in the EGS questionnaire among women with active employment-related fibromyalgia. A confidence level of 95% was used for the calculation.
  The sample will be divided into four groups, each comprising 40 women to account for a 15% anticipated dropout rate. The groups are as follows:
  Women with fibromyalgia who are actively working. Women with fibromyalgia on sick leave. Women with fibromyalgia with permanent work disability (officially recognized by the INSS).
  A control group of sedentary women without fibromyalgia
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Reliability of a Standardized Protocol for Functional Capacity Evaluation in Patients with Fibromyalgia | Baseline and 12 months
  The primary outcome will assess the reliability of a standardized protocol for evaluating the functional capacity of Spanish women with fibromyalgia. The protocol includes the Six-Minute Walk Test (6MWT), handgrip strength dynamometry, and the 8-foot Up & Go test. These measures will be evaluated for their consistency and accuracy in reflecting functional capacity over a 12-month period.
  For each test (6MWT, handgrip strength dynamometry and 8 feet up and go) the unit of measure for reliability will be intraclass correlation coefficient (ICC), measurement error (ME), small detectable change (SDC) and minimal important change (MIC).
Validity of a Standardized Protocol for Functional Capacity Evaluation in Patients with Fibromyalgia | Baseline and 12 months
  The primary outcome will assess the validity of a standardized protocol for evaluating the functional capacity of Spanish women with fibromyalgia. The protocol includes the Six-Minute Walk Test (6MWT), handgrip strength dynamometry, and the 8-foot Up & Go test. These measures will be evaluated for their consistency and accuracy in reflecting functional capacity over a 12-month period.
  For each test (6MWT, handgrip strength dynamometry and 8 feet up and go test) the unit of measure for validity will be correlation coefficient (r).

SECONDARY OUTCOMES:
Levels of Physical Activity (light, moderate and vigorous) and sedentary time in Different Fibromyalgia Patient Groups Measured by Triaxial Accelerometers | Baseline and 12 months
  This outcome will analyze the actual physical activity levels (light, moderate and vigorous) and sedentary time (min) of different patient groups with fibromyalgia-those who are working, those on sick leave, and those with recognized work disability-using triaxial accelerometers. The measure will assess differences in physical activity among these groups over a 12-month period.
Convergent Validity of Functional Assessments (6MWT, Handgrip Strength Dynamometry, and 8-Foot Up & Go) Compared to the Self-Administered Functional Impact Questionnaire (FIQ-R) | Baseline and 12 months
  This outcome will evaluate the convergent validity of the objective functional assessments-Six-Minute Walk Test (6MWT), handgrip strength dynamometry, and 8-Foot Up & Go test-by comparing them with the self-administered Functional Impact Questionnaire (FIQ-R). The aim is to determine how well these functional tests correlate with the FIQ-R
Predictive Validity of Functional Tests for Return to Work, Fibromyalgia Impact (FIQ-R), Short- and Medium-Term Quality of Life, Psychological Impact, and Social Impact | Baseline, 6 months, and 12 months
  This outcome will estimate the predictive validity of the functional tests (6MWT, handgrip strength dynamometry, and 8-Foot Up & Go) concerning several factors: return to work, fibromyalgia impact measured by the FIQ-R, short- and medium-term quality of life, psychological impact, and social impact. The aim is to assess how well these functional tests can predict these various outcomes over time. The unit of measure for predictive validity will be correlation coefficient.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - CAP Vila Olímpica, Barcelona, Barcelona
  - Facultat de Psicologia, Ciències de l'Educació i l'Esport (Blanquerna-URL), Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: No
Individual Patient Data (IPD) might not be shared due to concerns related to patient confidentiality and privacy. Given that the study involves sensitive health information, including details about fibromyalgia diagnosis, functional assessments, and personal health conditions, ensuring the protection of participants identities and data is crucial. Sharing IPD could potentially risk breaching patient confidentiality.
  Additionally, the study may have specific protocols or agreements in place that restrict the dissemination of individual data to protect participant privacy or comply with regulatory requirements. Ensuring proper data management and adhering to ethical standards for patient privacy and data protection are primary considerations that may impact the decision to share IPD.
  Therefore, while transparency is important, maintaining the confidentiality and security of individual patient data remains a priority.